CLINICAL TRIAL: NCT03410485
Title: Evaluation of the Combined Intraoperative Depth of Analgesia (NoL) and Depth of Anesthesia (BIS) Monitoring on the Patients' Recovery and Safety After Surgery: A Pilot Study
Brief Title: NoL and BIS Monitoring on Patients Recovery and Safety After Surgery
Acronym: CINAAMON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Canadian Anesthesiologists' Society (Other); Medasense Biometrics Ltd (Other)
Responsible Party: Principal Investigator, Philippe Richebé, Full Professor Anesthesiology, MD, PhD, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CER15083; CAS-2016-010 (Other Grant/Funding Number: Canadian Anesthesiologist Society)
Record Dates: First submitted 2016-10-11; First posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Pain; Anesthesia
Keywords: NoL index; Bispectral index; Intraoperative monitoring
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (C Group ) (Active Comparator): Intervention for intraoperative analgesic administration will be based on heart rate and blood pressure variations. Intervention for intraoperative hypnotice/desflurane administration will based on keeping the MAC at 0.8.
  Interventions: Device: Variation of baseline mean arterial pressure
- Monitoring (M Group ) (Experimental): Intervention for intraoperative analgesic administration will be based on the NOL index (to keep it below 25). Intervention for the desflurane administration will be based on the BIS index (to keep it between 40-60).
  Interventions: Device: BIS index/NoL index

INTERVENTIONS:
Device: BIS index/NoL index — Remifentanil i.v. infusion will be run between 0.03 and 0.15 mcg/kg/min and boluses (0.4mcg/kg) will be given to keep a NoL index between 10-20.
  Once intubated, the maintenance of anesthesia will be achieved with: desflurane set at 1 MAC to start, then adapted to the BIS between 45-55.
  Other Names: PMD200, Bispectral index
  Arms: Monitoring (M Group )
Device: Variation of baseline mean arterial pressure — Remifentanil i.v. infusion will be run between 0.03 and 0.15 mcg/kg/min and boluses (0.4mcg/kg) will be given to keep a baseline mean arterial pressure between 10% of variation.
  Once intubated, the maintenance of anesthesia will be achieved with: desflurane set at 1 MAC to start, then ajusted to 0.8 MAC.
  Arms: Control (C Group )

SUMMARY:
So far, only vital signs (mostly, blood pressure and heart rate) helped the anesthesiologist to administer hypnotic agents or analgesics. Many devices have offered pain monitoring for anesthetized patients, the most recent being the PMD200 device and its NoL index. The BIS index is widely used for depth of anesthesia monitoring. The hypothesis of this study is that the intraoperative combination of both the NoL and the BIS indices to guide the delivery of opioids and hypotonics respectively, will improve the quality of recovery as well as the safety after anesthesia in ERAS patients undergoing colonic surgery.

DETAILED DESCRIPTION:
Hypothesis is that the intraoperative use of the combination of 1) the NoL index (given by the PMD200TM monitor, Medasense LTD inc, Ramat, Israel) to monitor pain levels and to guide opioids' administration during surgery, and 2) the BIS index (Medtronic, St-Laurent, QC, Canada) to monitor the depth of hypnosis during anesthesia and to guide the administration of anesthetic halogenous gases, will improve the quality of recovery as well as the safety after anesthesia in ERAS (Early Rehabilitation After Surgery) patients undergoing colonic surgery under general anesthesia + epidural analgesia.

This study will compare a group of patients monitored by the classical monitoring (with anesthesia/analgesia guided by these classical parameters: heart rate, blood pressure; Control "C" group; no BIS, no NoL) to a group of patients monitored by the same classical monitoring implemented with the NoL/BIS indices (with analgesia/anesthesia guided by these 2 indices; Monitoring "M" group).

The primary objective of the study will be the total consumption of desflurane that is expected to be significantly reduced in the M group. Secondary objectives will be evaluating safety and side effects of anesthesia and opioids and we expect a reduction of the following parameters: time for awakening from anesthesia, time for extubation, time for transfer to PACU, intraoperative opioid consumption, opioid consumption in PACU and for 48h, time for readiness for discharge from PACU, incidence of adverse effects such as: nausea-vomiting / sedation / respiratory depression / itching / dizziness / cognitive dysfunction in PACU and for 48h, satisfaction of the patients at 24 and 48hs, pain scores at rest and at mobilization in PACU, at 24h and 48h. Quality of postoperative recovery after surgery and treatment satisfaction are also expected to be higher in the M group than in the C group.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I, II or III
* Patients aged 18 years
* Colo-rectal surgery
* Duration and type of surgery requiring an epidural analgesia via an epidural catheter placed prior the general anesthesia induction and an arterial line placed after induction of general anesthesia (classical management of ERAS program patients in our center)

Exclusion Criteria:

* chronic arhythmic condition
* chronic pain
* Adverse events prompting termination of protocol:
* Unexpected difficult airway requesting excessive, possibly painful airway manipulations.
* Unexpected surgical complications requiring strong haemodynamic support (transfusions, volume challenges, vasopressors, inotropic drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Total desflurane consumption | 10 hours
  Total consumption and absorption in ml/kg/h of desflurane in group C versus group M

SECONDARY OUTCOMES:
Hourly desflurane consumption | 10 hours
  Consumption and absorption of desflurane in ml/kg/h for each hour of surgery. These data are given by the Drager Perseus A500 ventilator per second during the surgery.
Total remifentanil consumption mcg/h | 10 hours
  Total consumption of i.v. remifentanil during surgery and for each hour of surgery
Hypotensive events | 10 hours
  Total number of hypotensive events during surgery defined as mean blood pressure below 10% of baseline
Total phenylephrine consumption mcg/h | 10 hours
  Total doses of intraoperative infused i.v. phenylephrine and doses per hour
Emergence time (seconds) | 30 min
  Time for awakening (eyes opening) at the end of the surgery, time for extubation, time for transfer to the PACU in seconds
Acute pain (NRS scores on scale from 0 to 10) | 48 hours postoperatively
  NRS scale pain score at rest
Analgesic requirement (total ml of epidural solution consumption) | 48 hours postoperatively
  cumulative dose over 48hs
Nausea and vomiting | 48 hours postoperatively
  on Nausea and vomiting scale from 0 to 4, cumulative scores over 48hours
Postoperative sedation | 48 hours postoperatively
  On POSS (postoperative sedation score) scale from 0 to 5, cumulative over 48 hours
Postoperative respiratory depression | 48 hours postoperatively
  yes or no (1 or 0) for 48 hours
PACU discharge time in minutes | 3 hours
  Time for readiness for PACU discharge based on Aldrete scores superior to 9.
Postoperative cognitive dysfunction | 5 days postoperatively
  Assessment of perioperative cognitive function using the classical MMSE scores over 5 days
Postoperative delirium | 5 days postoperatively
  Assessment of perioperative Delirium with NuDESC score over 5 days after surgery
Postoperative analgesia hydromorphone rescue | 5 days postoperatively
  Total hydromorphone rescue doses for 5 days, and total epidural doses in ml as continuous infusion + boluses (PCEA)
Recovery after surgery score on scale QOR15 (scale 0 to 150) | 5 days postoperatively
  Patients' perceived quality of recovery from anesthesia with QoR-15
Postoperative chronic pain (score 0 to 10) | 6 months postoperatively
  Presence and severity of persistent postoperative pain with DN4 questionnaires
Postoperative chronic pain (scale 0 to 60) | 6 months postoperatively
  Presence and severity of persistent postoperative pain SF-MPQ questionnaires
Mortality | 6 months postoperatively
  Rate of hospital mortality up to 6 months following surgery
Readmission | 6 months postoperatively
  Rate of hospital readmission up to 6 months following surgery
POCD/POD related inflammatory cytokines | 24h postoperatively
  Blood sample will be drawn and cytokines related to POCD/POD will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Richebé, Md, PhD, Principal Investigator — Full Professor
Locations (1):
- Hopital Maisonneuve Rosemont, CIUSSS de l'Est de l'Ile de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No